CLINICAL TRIAL: NCT03577717
Title: Efficacy of Computerized Cognitive Training in the Elderly With Mild Cognitive Impairment: Clinical Outcomes and Magnetoencephalographic Imaging
Brief Title: Efficacy of Computerized Cognitive Training in the Elderly With Mild Cognitive Impairment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was stopped due to time and budgetary constraints.
Sponsor: Taipei Hospital, Taiwan (Other)
Responsible Party: Principal Investigator, Wan-ying Chang, occupational therapist, Taipei Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201804
Record Dates: First submitted 2018-06-04; First posted 2018-07-05 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computerized cognitive training (Experimental): participants will be trained by the "Cookies for the brainy day", including memory, attention, calculation, executive functions, and language training.
  Interventions: Other: computerized cognitive training
- occupational therapy (Active Comparator): participants will receive craft activities of occupational therapy, such as weaving, origami etc.
  Interventions: Other: occupational therapy

INTERVENTIONS:
Other: computerized cognitive training — participants will be trained 30 minutes/day, 3 days/week for 4 consecutive weeks.
  Arms: computerized cognitive training
Other: occupational therapy — participants will receive craft activities of occupational therapy for 30 minutes/day, 3 days/week for 4 consecutive weeks.
  Arms: occupational therapy

SUMMARY:
Mild cognitive impairment (MCI) is the prodrome of the cognitive function declining before Alzheimer's disease or other dementia showed up, the impairments of language, visuospatial relationship, attention, and memory included and instrumental activities of daily living (IADL) influenced. MCI is considered as a transitional stage between normal aging and mild dementia, and the patients with MCI has differently fluctuated cognitive functions in a period of time, such as from normal cognition to MCI or developing to dementia. The annual conversion rate (ACR) of older adults with normal cognition developed to MCI is 30%, and 5% in clinical setting, and community, respectively. Not all of patients with MCI develop to Alzheimer's disease, the reversion of patients with MCI to normal cognition exists. However, MCI is a significant risk factor. The ACR of older adults with normal cognition or MCI developed to dementia is 1-2%, and 5-15%, respectively; moreover, about half of patients with MCI developed to dementia in 5 years.

Cognitive training (CT) improves cognitive functions with repetitive practicing standardized cognitive tasks of specific cognitive functions, such as memory, attention, or problem solving. CT has widely defined including strategy training, in which contained cognitive exercise, strategy indicating and practicing to reducing cognitive impairments and improving performances. CT is more effective for MCI. Recently, computer-based CT (CCT) with many advantages gradually replaced the traditional paper-pencil form. Brief systematic review showed that the computer-based intervention had positive effects on behavioral symptoms, such as depression and anxiety, in patients with MCI and/or dementia. Previous studies demonstrated that computer-based intervention exhibited moderate treatment effects on overall cognitive functions in patients with MCI, and also had positive effects on learning, short-term memory, and behavioral symptoms.

Older people with cognitive impairments is expected to increase by global aging. It is important for improving or maintaining cognitive functions of older adults with MCI. The efficacy of the CCT on cognitive functions, neuropsychiatric symptoms, daily functions, and brain activated imaging of the magnetoencephalography (MEG) of in older adults with MCI is worth to explore for busy clinical practice.

DETAILED DESCRIPTION:
The study design was a prospective and single-blinded randomized controlled trial. 36 participants with MCI were recruited and demographic data (age, gender, education level /years of education, marriage status etc.) were also collected. The MCI participants underwent the comprehensive review at baseline including neuropsychological assessment and Magnetic Resonance Imaging or Computerized Tomogram. Randomization treatment assignment will be generated by the random number table and assign the patient's intervention group accordingly. Sealed opaque envelopes containing the CCT group, or the dosage-matched control group sheets will be prepared and given to the therapists.

Based on the t-test effect size of index d 1.00 indicates, an estimated 17 participants in each group will be required for a power of 0.80 with a two-sided type I error of 0.05. Considering the 5% (q) drop rate, we will need to recruit 18 participants (N/1-q) for each group. The participants were randomly allocated to either the CCT group (18 participants) or the dosage-matched control group (18 participants) with individualized intervention for 30 minutes a day, 3 times a week for 4 consecutive weeks. Clinical outcome measures, and the imaging of the MEG were administered at pre- treatment, post-treatment and 1-month follow-up for further analysis.

Statistical analysis was performed using Statistical Package for the Social Sciences (SPSS) version 19.0. In statistical testing, two-sided p value ≤ 0.05 was considered statistically significant. The distributional properties of continuous variables were expressed by mean ± standard deviation (SD), categorical variables were presented by frequency and percentage. The differences in the distributions of continuous variables, categorical variables between the treatment and control groups were examined using two-sample t-test, Wilcoxon rank-sum test (or Mann-Whitney U test), and chi-square test. In addition, the minimum norm estimates (MNE), source-based time-frequency analysis, cross-frequency coupling, and functional connectivity were used to explore the differences of the activation of brain functions in participants between different treatment groups. The t-test was used to explore the differences of reaction time, rate of correction, and physical signals in stimulus reaction test of the MEG between in participants between different treatment groups. The correlation statistics was used to explore relationships between the scores of outcome measurements and the physical signals.

ELIGIBILITY:
Inclusion Criteria:

* (1) were aged ≥65 years
* (2) amnestic type MCI was made using National Institute on Aging-Alzheimer's Association workgroups diagnostic guidelines for Alzheimer's disease with the clinical dementia rating scale (CDR) global scores of 0.5
* (3) could follow command, understand the content of the assessments, and cooperate with treatment interventions through verbal communication

Exclusion Criteria:

* (1) had the score of Geriatric Depression Scale-Short Form (GDS-SF) > 7, indicating depression status
* (2) had the score of Barthel Index (BI)≠100, indicating dependent basic daily living of activities
* (3) were diagnosed with other MCI subtypes, including frontotemporal dementia or Lewy Body those present typically different MCI syndromes
* (4) had other neuropsychotic diseases
* (5) could not administrate with MEG
* (6) could not participate due to severe health problem

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Change scores of Quick Mild Cognitive Impairment screen | Baseline, 1 month, 2 months
  The Quick Mild Cognitive Impairment (Qmci) screen , a performance test, contains 6 subtests: Orientation, Registration, Clock Drawing, Delayed Recall, Verbal Fluency, and Logical Memory. The Qmci can be administered and scored in less than 5 min. The Qmci was validated with sound reliability and validity. The Qmci screen scores ranged from 0 to 100, with a higher score indicating greater cognitive function.
Change scores of Montreal Cognitive Assessment | Baseline, 1 month, 2 months
  The Montreal Cognitive Assessment (MoCA), a performance test, is a standardized and validated tool designed to measure cognitive functions in visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall, and orientation. The MoCA adds 1 score for those whose educational level ≤ 12 and scores ranged from 0 to 30, with a higher score indicating greater cognitive function.

SECONDARY OUTCOMES:
Change scores of Contextual Memory Test | Baseline, 1 month, 2 months
  The Contextual Memory Test is a standardized tool to measure the short-term and long-term retrospective memory and metacognition. The immediate and delayed memory is administrated by remembering 20 items related to daily context in 90 seconds. The scores of memory score, perceptual memory scores, and strategy-use scores were recorded.
Change scores of Color Trail Test | Baseline, 1 month, 2 months
  The Color Trail Test has A, and B parts. Participants needs to orderly connect randomized arrangement numbers in part A, and orderly and alternately connect randomized arrangement numbers in different colors in part B. The finished time and amounts of hint, miss, color miss, and near miss were recorded.
Change scores of Digits Span Tasks-forward and backward | Baseline, 1 month, 2 months
  The longest digits of forward and backward are 10 and 9, respectively. The total scores are 10 and 9, with a higher score indicating greater digit span memory.
Change scores of Cancellation Test | Baseline, 1 month, 2 months
  The Cancellation Test presents 10 Arabic numerals (0-9) for 30 digits per row (8 rows) with 2 target numerals (2, 8) in 45 seconds. The amounts of correction and miss were recorded.
Change scores of Pattern Comparison | Baseline, 1 month, 2 months
  The Pattern Comparisons presents 30 pairs of figures for distinguishing the same or not in 30 seconds. The amounts of correction, miss and total answers were recorded.
Change scores of Everyday Memory Questionnaire | Baseline, 1 month, 2 months
  Everyday Memory Questionnaire is a self-rated memory function questionnaire to reflect the frequency of memory miss in daily life. The frequency of memory miss, such as less than 1 time in 1-month, 2-3 times in 1-month, 1 time in 1 week, 2-6 times in 1 week, and more than 1 time in 1 day, in each situation scores ranged from 0 to 4 in 13 situations.
Change scores of Neuropsychiatric Inventory Questionnaire | Baseline, 1 month, 2 months
  The Neuropsychiatric Inventory Questionnaire (NPI-Q) measures symptoms severity and caregiver distress in 12 domains, such as apathy/indifference, appetite/eating problems, disinhibition, agitation/aggression, motor disturbance, anxiety, irritability, nighttime behaviors, depression/dysphoria, delusions, elation/euphoria, and hallucinations. The symptoms severity in each domain scores ranged from 1 to 3, with a higher score indicating more severe symptoms severity. In addition, the caregiver distress in each domain scores ranged from 0 to 5, with a higher score indicating more distress for caregiver.
Change scores of Brief University of California San Diego (UCSD) Performance-based Skills Assessment | Baseline, 1 month, 2 months
  The Brief University of California San Diego (UCSD) Performance-based Skills Assessment (UPSA-B) contains 2 aspects: financial skills, and communication skills. The UPSA-B can be administered and scored in 10-15 min and used to measure participants how to administrate daily activities and do it how well. The UPSA-B scores ranged from 0 to 100, with a higher score indicating greater daily function.
Change scores of Disability Assessment for Dementia Questionnaire (DAD) | Baseline, 1 month, 2 months
  The DAD contains 11 items of 3 domains: basic activity of daily living (dressing, hygiene, continence, eating), instrumental activity of daily living (meal preparation, telephoning, going on an outing, finance and correspondence, medications, and housework), and leisure activity (leisure). The scoring divides into 3 parts to measure about the initiation, planning and organization, and effective performance, and the scores of each part transforms to percentage for calculation. The higher percentage of each part indicates the less impairment in activities of daily living.

OTHER OUTCOMES:
Imaging change of the MEG | Baseline, 1 month, 2 months
  The 1-back working memory paradigm was used to explore the efficacy of each intervention. When one figure matches with the previous one, the participant needs to press the button for response as soon as possible. The Go-Nogo paradigm was to explore the reaction-inhibition functions. The participant needs to press the button for Go stimulus (1, 2, 4, 5, 6, 8, 9), and inhibits to press the button for Nogo stimulus (3, 7). Paired-stimulus paradigm is widely used for assessing the activation and inhibition functions of sensory cortex. The same of two stimuli (S1, S2) would show within 500 ms interval, and the magnitude of induced reaction of the second stimulus (S2) would be inhibited in normal physical condition. Calculating the S2/S1 ratio of paired-stimulus quantified the inhibition functions of sensory cortex, the much less ratio indicating the greater inhibition functions.

CONTACTS AND LOCATIONS:
Overall Officials: Wan-ying Chang, MS, Principal Investigator — Division of Occupational Therapy,Taipei Hospital, Ministry of Health and Welfare
Locations (1):
- Taipei Hospital, Ministry of Health and Welfare, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Data are available from the Institutional Review Board of the Taipei Hospital, Ministry of Health and Welfare for researchers who meet the criteria for access to confidential data.

REFERENCES:
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Bahar-Fuchs A, Clare L, Woods B. Cognitive training and cognitive rehabilitation for persons with mild to moderate dementia of the Alzheimer's or vascular type: a review. Alzheimers Res Ther. 2013 Aug 7;5(4):35. doi: 10.1186/alzrt189. eCollection 2013. PMID 23924584
- [Background] Barnes DE, Yaffe K, Belfor N, Jagust WJ, DeCarli C, Reed BR, Kramer JH. Computer-based cognitive training for mild cognitive impairment: results from a pilot randomized, controlled trial. Alzheimer Dis Assoc Disord. 2009 Jul-Sep;23(3):205-10. doi: 10.1097/WAD.0b013e31819c6137. PMID 19812460
- [Background] Bruscoli M, Lovestone S. Is MCI really just early dementia? A systematic review of conversion studies. Int Psychogeriatr. 2004 Jun;16(2):129-40. doi: 10.1017/s1041610204000092. PMID 15318760
- [Background] Caviness JN, Driver-Dunckley E, Connor DJ, Sabbagh MN, Hentz JG, Noble B, Evidente VG, Shill HA, Adler CH. Defining mild cognitive impairment in Parkinson's disease. Mov Disord. 2007 Jul 15;22(9):1272-7. doi: 10.1002/mds.21453. PMID 17415797
- [Background] Chen Y, Denny KG, Harvey D, Farias ST, Mungas D, DeCarli C, Beckett L. Progression from normal cognition to mild cognitive impairment in a diverse clinic-based and community-based elderly cohort. Alzheimers Dement. 2017 Apr;13(4):399-405. doi: 10.1016/j.jalz.2016.07.151. Epub 2016 Aug 30. PMID 27590706
- [Background] Cheng CH, Baillet S, Hsiao FJ, Lin YY. Effects of aging on neuromagnetic mismatch responses to pitch changes. Neurosci Lett. 2013 Jun 7;544:20-4. doi: 10.1016/j.neulet.2013.02.063. Epub 2013 Apr 2. PMID 23562510
- [Background] Cheng CH, Baillet S, Hsiao FJ, Lin YY. Effects of aging on the neuromagnetic mismatch detection to speech sounds. Biol Psychol. 2015 Jan;104:48-55. doi: 10.1016/j.biopsycho.2014.11.003. Epub 2014 Nov 15. PMID 25451380
- [Background] Cheng CH, Baillet S, Lin YY. Region-specific reduction of auditory sensory gating in older adults. Brain Cogn. 2015 Dec;101:64-72. doi: 10.1016/j.bandc.2015.10.004. Epub 2015 Oct 24. PMID 26507900
- [Background] Davis RN, Massman PJ, Doody RS. Cognitive intervention in Alzheimer disease: a randomized placebo-controlled study. Alzheimer Dis Assoc Disord. 2001 Jan-Mar;15(1):1-9. doi: 10.1097/00002093-200101000-00001. PMID 11236819
- [Background] De Vreese LP, Neri M, Fioravanti M, Belloi L, Zanetti O. Memory rehabilitation in Alzheimer's disease: a review of progress. Int J Geriatr Psychiatry. 2001 Aug;16(8):794-809. doi: 10.1002/gps.428. PMID 11536347
- [Background] Gaitan A, Garolera M, Cerulla N, Chico G, Rodriguez-Querol M, Canela-Soler J. Efficacy of an adjunctive computer-based cognitive training program in amnestic mild cognitive impairment and Alzheimer's disease: a single-blind, randomized clinical trial. Int J Geriatr Psychiatry. 2013 Jan;28(1):91-9. doi: 10.1002/gps.3794. Epub 2012 Apr 3. PMID 22473855
- [Background] Galante E, Venturini G, Fiaccadori C. Computer-based cognitive intervention for dementia: preliminary results of a randomized clinical trial. G Ital Med Lav Ergon. 2007 Jul-Sep;29(3 Suppl B):B26-32. PMID 18575355
- [Background] Gauthier S, Reisberg B, Zaudig M, Petersen RC, Ritchie K, Broich K, Belleville S, Brodaty H, Bennett D, Chertkow H, Cummings JL, de Leon M, Feldman H, Ganguli M, Hampel H, Scheltens P, Tierney MC, Whitehouse P, Winblad B; International Psychogeriatric Association Expert Conference on mild cognitive impairment. Mild cognitive impairment. Lancet. 2006 Apr 15;367(9518):1262-70. doi: 10.1016/S0140-6736(06)68542-5. PMID 16631882
- [Background] Garcia-Casal JA, Loizeau A, Csipke E, Franco-Martin M, Perea-Bartolome MV, Orrell M. Computer-based cognitive interventions for people living with dementia: a systematic literature review and meta-analysis. Aging Ment Health. 2017 May;21(5):454-467. doi: 10.1080/13607863.2015.1132677. Epub 2016 Jan 25. PMID 26806365
- [Background] Gelinas I, Gauthier L, McIntyre M, Gauthier S. Development of a functional measure for persons with Alzheimer's disease: the disability assessment for dementia. Am J Occup Ther. 1999 Sep-Oct;53(5):471-81. doi: 10.5014/ajot.53.5.471. PMID 10500855
- [Background] Gomar JJ, Harvey PD, Bobes-Bascaran MT, Davies P, Goldberg TE. Development and cross-validation of the UPSA short form for the performance-based functional assessment of patients with mild cognitive impairment and Alzheimer disease. Am J Geriatr Psychiatry. 2011 Nov;19(11):915-22. doi: 10.1097/JGP.0b013e3182011846. PMID 22024615
- [Background] Herrera C, Chambon C, Michel BF, Paban V, Alescio-Lautier B. Positive effects of computer-based cognitive training in adults with mild cognitive impairment. Neuropsychologia. 2012 Jul;50(8):1871-81. doi: 10.1016/j.neuropsychologia.2012.04.012. Epub 2012 Apr 21. PMID 22525705
- [Background] Hill NT, Mowszowski L, Naismith SL, Chadwick VL, Valenzuela M, Lampit A. Computerized Cognitive Training in Older Adults With Mild Cognitive Impairment or Dementia: A Systematic Review and Meta-Analysis. Am J Psychiatry. 2017 Apr 1;174(4):329-340. doi: 10.1176/appi.ajp.2016.16030360. Epub 2016 Nov 14. PMID 27838936
- [Background] Hughes TF, Flatt JD, Fu B, Butters MA, Chang CC, Ganguli M. Interactive video gaming compared with health education in older adults with mild cognitive impairment: a feasibility study. Int J Geriatr Psychiatry. 2014 Sep;29(9):890-8. doi: 10.1002/gps.4075. Epub 2014 Jan 22. PMID 24452845
- [Background] Huntley JD, Gould RL, Liu K, Smith M, Howard RJ. Do cognitive interventions improve general cognition in dementia? A meta-analysis and meta-regression. BMJ Open. 2015 Apr 2;5(4):e005247. doi: 10.1136/bmjopen-2014-005247. PMID 25838501
- [Background] Kaufer DI, Cummings JL, Ketchel P, Smith V, MacMillan A, Shelley T, Lopez OL, DeKosky ST. Validation of the NPI-Q, a brief clinical form of the Neuropsychiatric Inventory. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):233-9. doi: 10.1176/jnp.12.2.233. PMID 11001602
- [Background] Klimova B, Maresova P. Computer-Based Training Programs for Older People with Mild Cognitive Impairment and/or Dementia. Front Hum Neurosci. 2017 May 16;11:262. doi: 10.3389/fnhum.2017.00262. eCollection 2017. PMID 28559806
- [Background] Koepsell TD, Monsell SE. Reversion from mild cognitive impairment to normal or near-normal cognition: risk factors and prognosis. Neurology. 2012 Oct 9;79(15):1591-8. doi: 10.1212/WNL.0b013e31826e26b7. Epub 2012 Sep 26. PMID 23019264
- [Background] Lee GY, Yip CC, Yu EC, Man DW. Evaluation of a computer-assisted errorless learning-based memory training program for patients with early Alzheimer's disease in Hong Kong: a pilot study. Clin Interv Aging. 2013;8:623-33. doi: 10.2147/CIA.S45726. Epub 2013 Jun 7. PMID 23766638
- [Background] Lin F, Heffner KL, Ren P, Tivarus ME, Brasch J, Chen DG, Mapstone M, Porsteinsson AP, Tadin D. Cognitive and Neural Effects of Vision-Based Speed-of-Processing Training in Older Adults with Amnestic Mild Cognitive Impairment: A Pilot Study. J Am Geriatr Soc. 2016 Jun;64(6):1293-8. doi: 10.1111/jgs.14132. PMID 27321608
- [Background] Liu CY, Lu CH, Yu S, Yang YY. Correlations between scores on Chinese versions of long and short forms of the Geriatric Depression Scale among elderly Chinese. Psychol Rep. 1998 Feb;82(1):211-4. doi: 10.2466/pr0.1998.82.1.211. PMID 9520556
- [Background] Loewenstein DA, Acevedo A, Czaja SJ, Duara R. Cognitive rehabilitation of mildly impaired Alzheimer disease patients on cholinesterase inhibitors. Am J Geriatr Psychiatry. 2004 Jul-Aug;12(4):395-402. doi: 10.1176/appi.ajgp.12.4.395. PMID 15249277
- [Background] Manly JJ, Tang MX, Schupf N, Stern Y, Vonsattel JP, Mayeux R. Frequency and course of mild cognitive impairment in a multiethnic community. Ann Neurol. 2008 Apr;63(4):494-506. doi: 10.1002/ana.21326. PMID 18300306
- [Background] Mao HF, Kuo CA, Huang WN, Cummings JL, Hwang TJ. Values of the Minimal Clinically Important Difference for the Neuropsychiatric Inventory Questionnaire in Individuals with Dementia. J Am Geriatr Soc. 2015 Jul;63(7):1448-52. doi: 10.1111/jgs.13473. Epub 2015 Jun 5. PMID 26046666
- [Background] Mitchell AJ, Shiri-Feshki M. Rate of progression of mild cognitive impairment to dementia--meta-analysis of 41 robust inception cohort studies. Acta Psychiatr Scand. 2009 Apr;119(4):252-65. doi: 10.1111/j.1600-0447.2008.01326.x. Epub 2008 Feb 18. PMID 19236314
- [Background] Mok CC, Siu AM, Chan WC, Yeung KM, Pan PC, Li SW. Functional disabilities profile of chinese elderly people with Alzheimer's disease - a validation study on the chinese version of the disability assessment for dementia. Dement Geriatr Cogn Disord. 2005;20(2-3):112-9. doi: 10.1159/000086612. Epub 2005 Jun 30. PMID 15990425
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Neely AS, Vikstrom S, Josephsson S. Collaborative memory intervention in dementia: caregiver participation matters. Neuropsychol Rehabil. 2009 Oct;19(5):696-715. doi: 10.1080/09602010902719105. Epub 2009 Aug 21. PMID 19294562
- [Background] O'Caoimh R, Gao Y, McGlade C, Healy L, Gallagher P, Timmons S, Molloy DW. Comparison of the quick mild cognitive impairment (Qmci) screen and the SMMSE in screening for mild cognitive impairment. Age Ageing. 2012 Sep;41(5):624-9. doi: 10.1093/ageing/afs059. Epub 2012 May 18. PMID 22610464
- [Background] Petersen RC, Roberts RO, Knopman DS, Boeve BF, Geda YE, Ivnik RJ, Smith GE, Jack CR Jr. Mild cognitive impairment: ten years later. Arch Neurol. 2009 Dec;66(12):1447-55. doi: 10.1001/archneurol.2009.266. PMID 20008648
- [Background] Petersen RC, Smith GE, Waring SC, Ivnik RJ, Tangalos EG, Kokmen E. Mild cognitive impairment: clinical characterization and outcome. Arch Neurol. 1999 Mar;56(3):303-8. doi: 10.1001/archneur.56.3.303. PMID 10190820
- [Background] Quayhagen MP, Quayhagen M, Corbeil RR, Roth PA, Rodgers JA. A dyadic remediation program for care recipients with dementia. Nurs Res. 1995 May-Jun;44(3):153-9. PMID 7761291
- [Background] Rabipour S, Raz A. Training the brain: fact and fad in cognitive and behavioral remediation. Brain Cogn. 2012 Jul;79(2):159-79. doi: 10.1016/j.bandc.2012.02.006. Epub 2012 Mar 30. PMID 22463872
- [Background] Schafer KA, Tractenberg RE, Sano M, Mackell JA, Thomas RG, Gamst A, Thal LJ, Morris JC; Alzheimer's Disease Cooperative Study. Reliability of monitoring the clinical dementia rating in multicenter clinical trials. Alzheimer Dis Assoc Disord. 2004 Oct-Dec;18(4):219-22. PMID 15592134
- [Background] Spector A, Davies S, Woods B, Orrell M. Reality orientation for dementia: a systematic review of the evidence of effectiveness from randomized controlled trials. Gerontologist. 2000 Apr;40(2):206-12. doi: 10.1093/geront/40.2.206. PMID 10820923
- [Background] Spector A, Orrell M, Woods B. Cognitive Stimulation Therapy (CST): effects on different areas of cognitive function for people with dementia. Int J Geriatr Psychiatry. 2010 Dec;25(12):1253-8. doi: 10.1002/gps.2464. PMID 20069533
- [Background] Spector A, Thorgrimsen L, Woods B, Royan L, Davies S, Butterworth M, Orrell M. Efficacy of an evidence-based cognitive stimulation therapy programme for people with dementia: randomised controlled trial. Br J Psychiatry. 2003 Sep;183:248-54. doi: 10.1192/bjp.183.3.248. PMID 12948999
- [Background] Sun Y, Lee HJ, Yang SC, Chen TF, Lin KN, Lin CC, Wang PN, Tang LY, Chiu MJ. A nationwide survey of mild cognitive impairment and dementia, including very mild dementia, in Taiwan. PLoS One. 2014 Jun 18;9(6):e100303. doi: 10.1371/journal.pone.0100303. eCollection 2014. PMID 24940604
- [Background] Royle J, Lincoln NB. The Everyday Memory Questionnaire-revised: development of a 13-item scale. Disabil Rehabil. 2008;30(2):114-21. doi: 10.1080/09638280701223876. PMID 17852284
- [Background] Tarraga L, Boada M, Modinos G, Espinosa A, Diego S, Morera A, Guitart M, Balcells J, Lopez OL, Becker JT. A randomised pilot study to assess the efficacy of an interactive, multimedia tool of cognitive stimulation in Alzheimer's disease. J Neurol Neurosurg Psychiatry. 2006 Oct;77(10):1116-21. doi: 10.1136/jnnp.2005.086074. Epub 2006 Jul 4. PMID 16820420
- [Background] Tierney MC, Szalai JP, Snow WG, Fisher RH, Nores A, Nadon G, Dunn E, St George-Hyslop PH. Prediction of probable Alzheimer's disease in memory-impaired patients: A prospective longitudinal study. Neurology. 1996 Mar;46(3):661-5. doi: 10.1212/wnl.46.3.661. PMID 8618663
- [Background] Tsai CF, Lee WJ, Wang SJ, Shia BC, Nasreddine Z, Fuh JL. Psychometrics of the Montreal Cognitive Assessment (MoCA) and its subscales: validation of the Taiwanese version of the MoCA and an item response theory analysis. Int Psychogeriatr. 2012 Apr;24(4):651-8. doi: 10.1017/S1041610211002298. Epub 2011 Dec 12. PMID 22152127
- [Background] Tsai JC, Chen CW, Chu H, Yang HL, Chung MH, Liao YM, Chou KR. Comparing the Sensitivity, Specificity, and Predictive Values of the Montreal Cognitive Assessment and Mini-Mental State Examination When Screening People for Mild Cognitive Impairment and Dementia in Chinese Population. Arch Psychiatr Nurs. 2016 Aug;30(4):486-91. doi: 10.1016/j.apnu.2016.01.015. Epub 2016 Jan 21. PMID 27455923
- [Background] Valenzuela M, Sachdev PS. Harnessing brain and cognitive reserve for the prevention of dementia. Indian J Psychiatry. 2009 Jan;51 Suppl 1(Suppl1):S16-21. PMID 21416010
- [Background] Woods B, Aguirre E, Spector AE, Orrell M. Cognitive stimulation to improve cognitive functioning in people with dementia. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD005562. doi: 10.1002/14651858.CD005562.pub2. PMID 22336813
- [Background] Yoon JH, Lee JE, Yong SW, Moon SY, Lee PH. The mild cognitive impairment stage of dementia with Lewy bodies and Parkinson disease: a comparison of cognitive profiles. Alzheimer Dis Assoc Disord. 2014 Apr-Jun;28(2):151-5. doi: 10.1097/WAD.0000000000000007. PMID 24126215
- [Background] Yuill N, Hollis V. A systematic review of cognitive stimulation therapy for older adults with mild to moderate dementia: an occupational therapy perspective. Occup Ther Int. 2011 Dec;18(4):163-86. doi: 10.1002/oti.315. Epub 2011 Mar 21. PMID 21425381
- [Background] Gershon RC, Cella D, Fox NA, Havlik RJ, Hendrie HC, Wagster MV. Assessment of neurological and behavioural function: the NIH Toolbox. Lancet Neurol. 2010 Feb;9(2):138-9. doi: 10.1016/S1474-4422(09)70335-7. No abstract available. PMID 20129161
- [Background] Gershon RC, Wagster MV, Hendrie HC, Fox NA, Cook KF, Nowinski CJ. NIH toolbox for assessment of neurological and behavioral function. Neurology. 2013 Mar 12;80(11 Suppl 3):S2-6. doi: 10.1212/WNL.0b013e3182872e5f. PMID 23479538